CLINICAL TRIAL: NCT06095804
Title: A Single Center, Pilot Study to Evaluate the Feasibility of the Percutaneous Ultrasound Jejunostomy (PUJ)
Brief Title: Clinical Pilot Study of the Percutaneous Ultrasound Jejunostomy Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CoapTech (Industry)
Collaborators: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00107625
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Jejunostomy; Complications; Enteral and Supplement Feeds Adverse Reaction; Safety Issues
Keywords: Jejunostomy; Enteral Feeding; Long-term Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Percutaneous Ultrasound Jejunostomy (Experimental): Placement of a longterm jejunostomy tube using the PUMA-J System
  Interventions: Device: Percutaneous Ultrasound Jejunostomy

INTERVENTIONS:
Device: Percutaneous Ultrasound Jejunostomy — Placement of a jejunostomy tube using the PUMA-J System

SUMMARY:
The purpose of this study is to evaluate the feasibility and performance of the Percutaneous Ultrasound Jejunostomy (PUJ) procedure that utilizes a novel device (PUMA-J System) in conjunction with widely available ultrasound technology and endoscopic guidance.

The procedure will be performed in up to 10 eligible subjects. Patients will be followed for 2 days following performance of PUJ to assess for potential complications.

DETAILED DESCRIPTION:
Jejunostomy tubes (J-tubes) provide a path for nutrition delivery directly into the small intestinal lumen, bypassing the mouth, esophagus, and stomach for patients who have difficulty with proximal gut feeding. Many medical conditions may require J-tubes, including cancers, gastroparesis, and patients with high risk of aspiration.

A recent innovation by CoapTech addresses technical and procedural limitations of current jejunostomy tube placement methods by leveraging ultrasound for visualization and magnets for control of the jejunal loop. The Percutaneous Ultrasound Magnet Aligned (PUMA) System enables clinicians to affix jejunal loops superficially via magnetic coaptation and visualize the planned stomal tract using ultrasound. The purpose of this pilot clinical study is to test the feasibility of the PUMA-Jejunostomy (PUMA-J) System in adults requiring a jejunostomy tube.

This is a single-center, non-randomized, non-blinded feasibility study to evaluate the performance and safety of the PUJ procedure that utilizes a novel device (PUMA-J System).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained before any study-specific assessment is performed
* Male or female > 21 years of age
* Estimated tract length (skin to anterior abdominal wall) <= 4.5cm on prior imaging
* Indication for percutaneous jejunostomy tube placement determined to be present by the primary clinical care team (examples below):

  * High aspiration risk
  * Malnourished- chronically ill and/or neurologically impaired requiring jejunal feeding for >30 Days.
  * Neoplasia (stomach and esophagus)
  * Gastric and duodenal obstruction
  * Gastrointestinal dysmotility (gastroparesis)
  * Altered anatomy (gastric-esophageal surgeries)
  * Other indication deemed to be appropriate by the study team
* Patient determined to be an appropriate candidate for percutaneous jejunostomy by the study team
* Women of childbearing potential must have negative serum or urine pregnancy test during the current hospitalization

Exclusion Criteria:

* Temperature ≥ 38 C
* Systolic BP < 90 or > 180 mmHg
* Heart Rate < 50 or > 120
* Presence of a contraindication to being in proximity to a magnet (e.g. pacemaker)
* History of prior major abdominal surgery
* Patients with HgB < 7g/dL, or fluid resuscitated within 48hrs prior, or history of life-threatening gastrointestinal bleeding within 1 month
* Pregnant or nursing (lactating) women
* Involvement in other investigational trials within 30 days prior to screening
* Absolute contraindications:

  * Sepsis
  * Severe ascites
  * Peritonitis
  * Coagulopathy (international normalized ratio (INR) greater than 1.5 or a platelet count of less than 50,000/uL)
  * Abdominal wall infection at the site of planned tube insertion
  * Interposed organs as determined by imaging
  * Abnormal upper gastrointestinal anatomy (e.g., partial or Total gastrectomy, Esophageal strictures)
  * Inflammatory, or infiltrative diseases of the small bowel and/or anterior abdominal wall.
  * Other standard general contraindications to endoscopy
  * Pacemakers or other electronically active implantable devices
  * Small bowel fistula
* Any other medical condition(s) that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Procedure timeframe
  Rate of procedural success in completing jejunostomy tube placement using the PUMA-J System

SECONDARY OUTCOMES:
Procedural Aborts | Procedure timeframe
  Description of occurrences of procedure abort
Device Related Serious Adverse Events | 48 hours of procedure performance
  Rate of Device Related Adverse Events following Jejunostomy procedure
Adverse Events | 48 hours of procedure performance
  Rate of all Adverse Events following Jejunostomy procedure
Rate of inadvertent puncture of vital organs | Procedure timeframe
  Description of occurrences of inadvertent puncture of vital organs during performance of procedure
Requirement for salvage surgery due to complication of the procedure | 48 hours of procedure performance
  Description of occurrences of salvage surgery performed due to complication of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No